CLINICAL TRIAL: NCT03807401
Title: To Simulate Prismatic Adaptation in Healthy Subject : a Technical Innovation in Favour of Autonomy and Independence in Daily Life Following a Brain Injury
Brief Title: A Technical Innovation of Prismatic Adaptation Test in Healthy Subject, in Favour of Autonomy and Independence in Daily Life Following a Brain Injury
Acronym: PRIS'TUEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0721; 2018-A03175-50 (Other: ID-RCB)
Record Dates: First submitted 2018-11-27; First posted 2019-01-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Virtual Reality; prismatic adaptation; motor imagery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical prismatic adaptation (Active Comparator): Classical prismatic adaptation arm will be divided into two subgroups corresponding to the side of the prismatic displacement (right or left)
  Interventions: Behavioral: Prismatic goggles
- Virtual prismatic adaptation (Experimental): virtual prismatic adaptation arm will be divided into two subgroups corresponding to the side of the prismatic displacement (right or left)
  Interventions: Behavioral: Virtual reality device
- Imaged prismatic adaptation (Experimental): Imaged prismatic adaptation arm will be divided into two subgroups corresponding to the side of the prismatic displacement (right or left)
  Interventions: Behavioral: Prismatic goggles

INTERVENTIONS:
Behavioral: Prismatic goggles — Goggles inducing a lateral displacement of the virtual field of ten degrees. Participants will be asked to wear those goggles during adaptation session and to perform pointing movement toward visual target.
  Arms: Classical prismatic adaptation
Behavioral: Virtual reality device — The lateral displacement will be simulated thanks to a virtual reality environment. Participants will wear an Oculus Rift instead of the prismatic goggles and will perform pointing movement as well.
  Arms: Virtual prismatic adaptation
Behavioral: Prismatic goggles — Goggles inducing a lateral displacement of the virtual field of ten degrees. Participants will be asked to wear those goggles during adaptation session and to mentally perform pointing movement toward visual target. There will be no concurrent movement execution.
  Arms: Imaged prismatic adaptation

SUMMARY:
Unilateral neglect is a neuropsychological disorder reflected by a disturbance in the spatial exploration and distribution of directed attention affecting the contralateral part of space and body relatively to the brain lesion. The chronic aspect of this pathology leads to a poor progression following rehabilitation and a decreased independence of patients in daily life. Thus, it is necessary to set up efficient and long lasting therapies for unilateral neglect patients to improve their daily quality of life. Prismatic adaptation is now a classical method which allows patients to improve their neglect through corrective pointing movements in response to a lateral displacement of the visual field. A large and growing body of literature has investigated prismatic adaptation as a very promising rehabilitation method, improving both visuomotor and cognitive features of unilateral neglect. However, its effects are somehow irregular and clinical applications of this method are still limited. The necessity for patients to come to the hospital to take advantage of prismatic adaption sessions draws some limitations about our knowledge concerning 1) the temporal dynamic of prism adaptation effects on a long-term basis and 2) the optimal duration of treatment (most of the time constrained by the hospitalization duration) and its therapeutical effects on a very long-term basis. Moreover, a large number of patients also suffer from motor deficits which reduce the possibility to optimize the prismatic adaptation session.

Thus, the aim of this project is to develop and validate others modalities of prismatic adaptation which can be applied at home and for a longer duration. These modalities should allow the investigator to get insights about the temporal dynamic of prismatic adaptation on the cognitive system. First, the investigator will investigate the effects of a prismatic adaptation modality using virtual reality to reproduce the lateral displacement induced by the prismatic goggles. He will also investigate prismatic adaptation induced by motor imagery, i.e. with mental representations of pointing movements without concomitant motor execution. This project could enhance the fundamental knowledge and enable to design new modalities of therapeutical use of prismatic adaptation (virtual or imaged) so as to allow a home-based treatment and follow-up. Thus, the aim of this project is to demonstrate the implication of similar mechanisms through different modalities (virtual and imaged compared to classical application) and the feasibility of these new modalities of healthy subjects. Thereafter, the aim will be to use knowledge acquired during this project to set up clinical trials to test for the efficiency of these modalities on a long-term basis in a pathological population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Right-handed
* Aged 18 to 70
* Normal or corrected vision
* Signed written informed consent
* Affiliated to a health care organism.

Exclusion Criteria:

* Neurological or psychiatric disorder
* Cognitive disorders
* presence of corrective eyeglasses
* Right upper limb orthopedic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
sensorimotor performances : measure of deviations in mm | Day 0 - right before adaption
  Task 1 : Line bisection to assess visuo-spatial bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Line bisection test, the reference point is the middle of the line.
Visuospatial performances : measure of deviations in mm | Day 0 - right before adaption
  Task 1 : Line bisection to assess visuo-spatial bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Line bisection test, the reference point is the middle of the line.
Visuospatial performances : measure of deviations in mm | Day 0 - right after adaption
  Task 1 : Line bisection to assess visuo-spatial bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Line bisection test, the reference point is the middle of the line.
sensorimotor performances : measure of deviations in mm | Day 0 - right after adaption
  Task 1 : Line bisection to assess visuo-spatial bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Line bisection test, the reference point is the middle of the line.
Visuospatial performances : measure of deviations in mm | Day 0 - right before adaption
  Task 2 : Goal-directed pointing to assess sensorimotor bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Goal-directed pointing test, the reference point is the target.
sensorimotor performances : measure of deviations in mm | Day 0 - right before adaption
  Task 2 : Goal-directed pointing to assess sensorimotor bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Goal-directed pointing test, the reference point is the target.
Visuospatial performances : measure of deviations in mm | Day 0 - right after adaption
  Task 2 : Goal-directed pointing to assess sensorimotor bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Goal-directed pointing test, the reference point is the target.
sensorimotor performances : measure of deviations in mm | Day 0 - right after adaption
  Task 2 : Goal-directed pointing to assess sensorimotor bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Goal-directed pointing test, the reference point is the target.
Visuospatial performances : measure of deviations in mm | Day 0 - right before adaption
  Task 3 : Straight Ahead pointing to assess proprioceptive bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Straight Ahead pointing and Visual judgement tests, the reference point is a central imaginary line
sensorimotor performances : measure of deviations in mm | Day 0 - right before adaption
  Task 3 : Straight Ahead pointing to assess proprioceptive bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Straight Ahead pointing and Visual judgement tests, the reference point is a central imaginary line
Visuospatial performances : measure of deviations in mm | Day 0 - right after adaption
  Task 3 : Straight Ahead pointing to assess proprioceptive bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Straight Ahead pointing and Visual judgement tests, the reference point is a central imaginary line
sensorimotor performances : measure of deviations in mm | Day 0 - right after adaption
  Task 3 : Straight Ahead pointing to assess proprioceptive bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
  For the Straight Ahead pointing and Visual judgement tests, the reference point is a central imaginary line
Visuospatial performances : measure of deviations in mm | Day 0 - right before adaption
  Task 4 : Visual judgement to assess visual bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
sensorimotor performances : measure of deviations in mm | Day 0 - right before adaption
  Task 4 : Visual judgement to assess visual bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
Visuospatial performances : measure of deviations in mm | Day 0 - right after adaption
  Task 4 : Visual judgement to assess visual bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.
sensorimotor performances : measure of deviations in mm | Day 0 - right after adaption
  Task 4 : Visual judgement to assess visual bias In the test, the investigator will measure the deviation (in mm) between the response of the subject and the reference point.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROSSETTI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Lyon Neuroscience Research Center, Bron, France